CLINICAL TRIAL: NCT01736527
Title: Tear Fluid Levels of Loteprednol Etabonate Ophthalmic Gel 0.5% at 6, 9, 12, and 24 Hours Following a Single Instillation in Healthy Volunteers
Brief Title: Tear Fluid Levels of Loteprednol Etabonate Ophthalmic Gel 0.5% Following a Single Instillation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 808
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-08

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Loteprednol Etabonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LE Gel (Experimental): A single dose LE Gel 0.5% administered into the study eye, tear samples collected at 6, 9, 12, and 24 hours after instillation by Schirmer strip to measures levels of LE in tears.
  Interventions: Drug: LE Gel

INTERVENTIONS:
Drug: LE Gel — Single drop of LE Gel 0.5% administered to the study eye on visit 2
  Other Names: Lotemax

SUMMARY:
To assess the levels of loteprednol etabonate (LE) in tear fluid following a single topical instillation of LE ophthalmic gel 0.5% formulation to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy volunteers with physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Subjects must have a best-corrected visual acuity of 20/20 or better in each eye.
* Subjects must have no active ocular disease or allergic conjunctivitis.
* Subjects must have a Schirmer test (without anesthesia) of ≥ 10mm in 5 minutes.
* Subjects must not be using any topical ocular medications or systemic medication other than acetaminophen.
* Male subjects or female subjects who are not of childbearing potential. Female subjects are considered to not be of childbearing potential if they are postmenopausal for at least 12 months or permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy)

Exclusion Criteria:

* Subjects having an intraocular pressure less than 5 mmHg or greater than 22 mmHg or any type of glaucoma.
* Subjects with a history of ocular trauma, infection, or inflammation within the last 3 months.
* Subjects having any contraindication to the use of, or known sensitivity or allergy to, the study drug(s) or their components.
* Subjects wearing contact lenses on the day of Visit 2 and/or Visit 3 of the study
* Subjects having, at the Investigator's discretion, the presence of any significant illness that could be expected to interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Schafer, OD, MS, Principal Investigator — Bausch & Lomb Incorporated; Raphaele Siou Mermet, MD, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Research Clinic, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center, open label, single dose study in healthy volunteers. First participant enrolled 01/08/2013, last participant exited: 01/18/2013.
Pre-assignment Details: A total of 17 participants were screened for this study. Of those screened, 12 participants were included to receive treatment; these subjects constituted the Safety population. No participants discontinued from the study.
Groups:
- LE Gel: A single dose LE Gel 0.5% administered into the study eye, tear samples collected at 6, 9, 12, and 24 hours after instillation by Schirmer strip to measures levels of LE in tears.
  LE Gel : Single drop of LE Gel 0.5% administered to the study eye on visit 2
Period: Overall Study
Arm/Group | LE Gel
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LE Gel
Number analyzed (Participants) | 12
Age, Customized [Mean (Standard Deviation); unit: years] | 45.6 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Tear Fluid Levels
Description: Following a single dose of LE gel 0.5% administered into the study eye, tear samples will be collected via a Schirmer strip at 6, 9, 12 and 24 hours following the dose
Time Frame: 6 hours
Population: The primary analysis includes all subjects in the safety population with tear samples collected within the corresponding time window.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | LE Gel
Number analyzed (Participants) | 12
μg/g | 113.633 (116.0133)

2. Primary Outcome: Tear Fluid Levels
Description: as for outcome 1
Time Frame: 9 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | LE Gel
Number analyzed (Participants) | 10
μg/g | 19.667 (18.1625)

3. Primary Outcome: Tear Fluid Levels
Description: as for outcome 1
Time Frame: 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | LE Gel
Number analyzed (Participants) | 12
μg/g | 26.877 (29.6464)

4. Primary Outcome: Tear Fluid Levels
Description: as for outcome 1
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | LE Gel
Number analyzed (Participants) | 11
μg/g | 2.408 (3.3631)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: All 12 subjects were exposed to a single dose of LE Gel.
Arm/Group | LE Gel
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LE Gel (N=12)
Headache (Nervous system disorders) | 1 (1) — Non-Ocular Treatment-Emergent Adverse Events Population: Safety

LIMITATIONS AND CAVEATS:
All 12 subjects were exposed to a single dose of LE Gel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes